CLINICAL TRIAL: NCT07314437
Title: Randomised Trial (With Integrated Pilot) Evaluating Whether a Standardised Approach, Educational Package (Including Checklist) Improve Recognition of Major Life-threatening Injuries in the Hot Reporting of Trauma Scans
Brief Title: 5 Minute 'HOT' Trauma CT Rates Of Detection Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Principal Investigator, Paul Jenkins, Consultant Interventional Radiologist, University Hospital Plymouth NHS Trust
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: 25/RAD/176; 361877 (Other: Integrated Research Application System); 70122 (Other: Central Portfolio Management System)
Record Dates: First submitted 2025-11-25; First posted 2026-01-02 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Trauma (Including Fractures); Trauma Abdomen; Trauma Blunt; Trauma Centers
Keywords: Trauma; CT; Hot Report; Radiology; HOT-RODs
MeSH Terms: conditions — Wounds and Injuries; Abdominal Injuries; Wounds, Nonpenetrating | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The primary analysis will be comparative between the pickup rate between the first and second imaging set within groups 1 and 2. Group 3 will act a control group to determine the effect of repetition on skill development rather than the education package. Subgroup analysis of clinicians by demographics including trauma experience will be performed.
Who Masked: Participant
Masking Description: Each Group will not be aware of the intervention or education or content the other Group receives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 3 Control Group (No Intervention): No intervention. Control Group.
- Group 1 Intervention Group A Images (Experimental): Group 1 will report image bank A, receive the educational intervention and then report image bank B with the checklist.
  Interventions: Other: Education
- Group 2 Intervention Group B Images (Experimental): Group 2 will report image bank B, receive the educational intervention and then report image bank A.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — The three groups will report 2 image banks of 15 CT images each. Image bank A will contain 15 CT images each with a brief history including the mechanism of injury. Image bank B will contain 10 new CT images and 5 CT images contained within image bank A, but with an altered but compatible mechanism of injury.
  Group 1 will report image bank A, receive the educational intervention and then report image bank B with the checklist. Group 2 will report image bank B, receive the educational intervention and then report image bank A. Group 3 will report image bank A and B without any intervention.
  Arms: Group 1 Intervention Group A Images; Group 2 Intervention Group B Images

SUMMARY:
Many injured patients receive urgent CT imaging to identify major injury. CT imaging of trauma patients is often time critical and the accurate detection of life-threatening findings on this CT is essential. Often following a scan a radiologist is not immediately available to review the imaging, however other members of the trauma team have access to the imaging and may be in a position to provide a "hot" report. In this study we aim to demonstrate if an educational intervention with a checklist improves accuracy of the hot report.

DETAILED DESCRIPTION:
This is a randomised controlled trial to evaluate whether a standardised approach, educational package (with checklist) may improve recognition of major life-threatening injuries in the hot reporting of trauma scans. A pilot study with 20 participants allocated to the two groups on 1:1 ratio which will receive the education package, will inform feasibility of the larger study.

The larger study will recruit 300 participants, 100 on each group on 1:1:1 ratio, to evaluate the primary objective.

Participants will be clinicians who volunteer to participate in an online educational package. Participant data will be collected by the online platform under a unique identifier. Results will then be extracted from the platform and then associated with the demographic data on the trust system.

Following application of inclusion and exclusion criteria, participants will be allocated into one of three groups, and assigned a participant number. The test data set will consist of cases that have been pseudo anonymised with the key stored on trust systems.

ELIGIBILITY:
Inclusion Criteria:

* Medical professionals involved in trauma image review.
* This includes clinicians who are emergency department doctors, radiologists and other specialties.
* Non-radiologist clinicians will be participating completing the hot reports, radiologists will be evaluating their submissions and assessing their accuracy.

Exclusion Criteria:

* Unable to review CT imaging due to lack of previous experience or disability that prevents them from doing so.
* Under 18 years old.
* Not a medical professional or clinician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Rates of detection and error of a hot CT report. | 1 year
  Measure using percentage difference in hot report accuracy rates between those who receive the educational package and those who did not. Participants will submit their answers onto the platform and these will be evaluated by Radiologists familiar with the trauma scans the participants have reviewed. The primary analysis will be comparative between the pickup rate between the first and second imaging set within groups 1 and 2. Group 3 will act a control group to determine the effect of repetition on skill development rather than the education package.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Plymouth, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We aim to make IPD available after the project's 1st publication with the data analysed. We anticipate that this will be a maximum of one year following the anticipated completion date of the project, 15th January 2028.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The IPD and supporting information will be made available via the request process outlined below after the project's first publication with the data analysed. We anticipate this will be a maximum of one year following the anticipated completion date of the study (15th January 2027).
Access Criteria: Requests for data sharing can be made after publication of the primary results paper. Requests should be made to the Chief Investigator in the first instance. Requesters will be asked to complete an application form detailing specific requirements, rationale, and proposed usage. The CI and study sponsor (including the sponsor's Research Governance Manager (or deputy), the Information Governance Team, Calidcott Guardian, IM&T Security Officer and the researcher funder, as appropriate) will review all requests.
  Consideration will be given to:
  1. The viability and suitability of the request
  2. Appropriate steps have been taken to minimise the risk of identifying participants
  3. Data security policies and procedures of recipient organisation (including country if abroad) and other regulatory requirements are applicable
  4. The credentials of the requestor
  Where access to requested data is granted, requesters organisation must sign a data sharing agreement before they can access any